CLINICAL TRIAL: NCT03140917
Title: Multimodal Assessment of Liver Volume and Function in Patients With Colorectal Liver Metastases
Brief Title: Multimodal Assessment of Liver Volume and Function
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Ernesto Sparrelid, MD PhD, Karolinska University Hospital
Other Study IDs: Liver fx study
Record Dates: First submitted 2017-04-28; First posted 2017-05-04 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: Liver function; Future liver remnant; Chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multimodal liver function assessment — HBS, MRI, CE-CT and ICG

SUMMARY:
In liver surgery peroperative assessment och the future liver remnant (FLR) is pivotal in order to avoid posthepatectomy liver failure. To date this is mainly performed by measuring the volume of the FLR. Of course FLR volume acts as a surrogate measure of FLR function and the correlation between volume and function is not always accurate. Several techniques to assess FLR function has been proposed. Hepatobiliary scintigraphy (HBS) and Dynamic MRI are the two such methods. In this study we compare HBS and MRI, in addition to contrast-enhanced CT and ICG, repeatedly performed before and after right hepatectomy in patients with colorectal liver metastases treated with neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* CRLM treated with neoadjuvant chemotherapy subjected to right hepatectomy

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CRLM treated with neoadjuvant chemotherapy subjected to right hepatectomy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Correlation between HBS and MRI in assessment of FLR function preop | Preop
  HBS, MRI, CT and ICG performed the day before surgery

SECONDARY OUTCOMES:
Correlation between HBS and MRI in assessment of FLR function POD 7 | POD 7
  HBS, MRI, CT and ICG performed 7 days after surgery
Correlation between HBS and MRI in assessment of FLR function POD 28 | POD 28
  HBS, MRI, CT and ICG performed 28 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Nilsson, MD PhD, Study Chair — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No